CLINICAL TRIAL: NCT06538935
Title: A Phase II, Open-label, Two Arm, Investigator-initiated Trail of Stereotactic Radiotherapy (SBRT) in Combination With an Anti-PD-L1 Inhibitor Adbelimumab and Apatinib for Perioperative and Conversion Therapy of Hepatocellular Carcinoma
Brief Title: SBRT Combined With Adbelimumab and Apatinib for Perioperative and Conversion Therapy of Hepatocellular Carcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCC
Record Dates: First submitted 2024-07-31; First posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-07

CONDITIONS: Hepatocellular Carcinoma; SBRT; Immune Checkpoint Blockade; Tyrosine Kinase Inhibitor
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Perioperative queue (Experimental): SBRT: SBRT: 8-30Gy/1-6F（dose is determined according to the tumor diameter）； Adbelimumab: 2-3 cycles of neoadjuvant therapy before surgery, 1200mg iv d1 q3w; Apatinib : D1-D21 : 250 mg, orally, qd; Before surgery, the patient's surgical pathology samples still need to be collected.
  After surgery, patients would receive Adbelimumab and Apatinib as adjuvant therapy .No more than 17 cycles before and after surgery.
  Interventions: Drug: adbelimumab; Procedure: SBRT; Drug: apatinib
- Conversion queue (Experimental): SBRT: tumor thrombus dose 30Gy /5-6F; Primary tumor dose is referred to Perioperative queue; Adbelimumab: 1200mg iv d1 q3w; Apatinib : D1-D21 : 250 mg, orally, qd; Treatment continues till PD,death,intolerable toxicity,or meet the criteria for Successful transformation(the maximum duration of adbelizumab combined with Apatinib conversion therapy was 1 year).
  Interventions: Drug: adbelimumab; Procedure: SBRT; Drug: apatinib

INTERVENTIONS:
Drug: adbelimumab — adbelimumab：1200mg iv d1 q3w
Procedure: SBRT — SBRT: SBRT: 8-30Gy/1-6F（dose is determined according to the tumor diameter）; tumor thrombus dose 30Gy /5-6F;
Drug: apatinib — apatinib：250mg po, qd

SUMMARY:
This is a Phase II , Open-label , Investigator-initiated Trail of SBRT in Combination With Adbelimumab and Apatinib in Patients With Hepatocellular Carcinoma(HCC).This study aims to evaluate the safety and efficacy of SBRT in Combination With Adbelimumab and Apatinib as a preoperative and conversion treatment of HCC.

DETAILED DESCRIPTION:
This is an Open, Two Arm, Exploratory and Phase II Clinical Trial of SBRT Combined With Adbelimumab (an Anti-PD-L1 Inhibitor) and Apatinib in Patients With Hepatocellular Carcinoma(HCC) as Perioperative and Conversion Treatment. we conduct this study in order to observe and evaluate the efficacy and safety of SBRT Combined With Adbelimumab and Apatinib in treatment of patients with HCC. Primary Efficacy Endpoint: Perioperative cohort-Pathological complete response Rate (pCR); Conversion cohort-Objective Response(ORR) (According to RECIST Version 1.1).Secondary Efficacy Endpoints:Perioperative cohort-Major pathologic response (MPR) ,Event-free survival (EFS) and Overall survival (OS )；Conversion cohort-Radical (R0) resection rate,Disease control rate (DCR),Progression free survival(PFS) and Overall survival (OS ).Safety and tolerance will be evaluated by incidence, severity and outcomes of AEs.

ELIGIBILITY:
Inclusion Criteria:

1. The patient volunteered to participate in the study and signed an informed consent form
2. ≥18 years of age，Male or female
3. Subjects are diagnosed with histologically or cytologically confirmed HCC
4. Subjects haven't received any systemic treatment for HCC before admission.
5. Subjects enrolled must have measurable lesion(s) according to the RECIST 1.1 standard
6. ECOG performance status of 0 or 1
7. Life expectancy ≥ 12 weeks
8. Subjects are diagnosed with resectable stage IB- IIIA HCC cancer.
9. The main organ's function is normal and it should meet the following criteria(Excludes use of any blood components and cell growth factors during the screening period)

   * Absolute neutrophil count≥1.5×109 /L
   * Platelets≥75×109/L ;Hemoglobin≥9.0 g/dL; Serum albumin≥3g/dL
   * Thyroid stimulating hormone (TSH)≤1.0×upper limit of normal(ULN)（If abnormal, T3 and T4 levels should be examined at the same time）
   * Total bilirubin (TBIL)≤1.5×upper limit of normal (ULN); ALT and AST≤1.5×upper limit of normal(ULN); AKP≤ 2.5×upper limit of normal(ULN)
   * Serum creatinine ≤1.5×ULN or creatinine clearance > 60 mL/minute (using Cockcroft-Gault formula)

Exclusion Criteria:

1. Known hepatocholangiocarcinoma, sarcomatoid HCC, mixed cell carcinoma and lamellar cell carcinoma; other active malignant tumor except HCC within 5 years or simultaneously
2. Be ready for or previously received organ or allogenic bone marrow transplantation
3. Moderate-to-severe ascites with clinical symptoms
4. History of gastrointestinal hemorrhage within 6 months prior to the start of study treatment or clear tendency of gastrointestinal hemorrhage.
5. Abdominal fistula, gastrointestinal perforation or intraperitoneal abscess within 6 months prior to the start of study treatment.
6. Known genetic or acquired hemorrhage or thrombotic tendency.
7. Thrombosis or thromboembolic event within 6 months prior to the start of study treatment.
8. Cardiac clinical symptom or disease that is not well controlled.
9. Subjects have uncontrollable hypertension (systolic pressure ≥ 140 mmHg or diastolic pressure ≥ 90 mmHg), despite patients have taken the best drug treatment ；Subjects have had a hypertensive crisis or hypertensive encephalopathy
10. Patient develops severe vascular disease within 6 months before the start of study treatment.
11. Patients with severe, unhealed or split wounds and active ulcers or untreated fractures.
12. Patients who underwent surgical treatment within 4 weeks prior to the start of study treatment.
13. Factors to affect oral administration (such as patients unable to swallow oral medications, malabsorption syndrome etc. situations evidently affect drug absorption).
14. Patients with gastrointestinal diseases such as intestinal obstruction (including incomplete intestinal obstruction) or those who may have caused gastrointestinal bleeding, perforation or obstruction.
15. There is evidence of intragastric gas that cannot be explained by puncture or recent surgery.
16. Previous or current presence of metastasis to central nervous system.
17. Subjects have history of hepatic encephalopathy.
18. The subject has an interstitial lung disease that is symptomatic or may interfere with the discovery or management of suspected drug-related lung toxicity; previous and current subjects with a history of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, drug-associated pneumonia, severe impaired lung function, etc.
19. The patient has any active autoimmune disease or a history of autoimmune disease expected relapse.
20. Severe infection within 4 weeks prior to the start of study treatment.
21. A history of immunodeficiency, including HIV-positive or other acquired, congenital immunodeficiency disease.
22. The patient is pregnant or breastfeeding.
23. Subjects were vaccinated with live attenuated vaccine within 28 days before the first dose or expected to receive this vaccine within 60 days after the last dose or during the study period.
24. Treatment of other investigational product(s) within 28 days prior to the start of study treatment.
25. Other factors deemed unsuitable for participation in this study by the researchers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response Rate (Perioperative cohort) | 4 months
  No histologic evidence of malignancy or only the ingredients of carcinoma in situ was found in primary tumors
Objective Response (Conversion cohort) | 12 months
  It is defined as the proportion of patients whose tumors shrink to a predetermined size and maintain a minimum time limit. It includes the cases of CR and PR.

SECONDARY OUTCOMES:
Event-free survival | 5 year
  Refers to the time from the start of the group to the occurrence of any event
Major pathologic response | 4 months
  It is defined as residual tumors less than 10% after neo-adjuvant therapy
Overall survival | 5 year
  It is defined as the time from randomization to death from any cause during the course of the study
Safety as measured by the rate of AEs | 1 month
  Safety will be evaluated by incidence, severity and outcomes of adverse events (AEs)